CLINICAL TRIAL: NCT06773910
Title: An Open-label, Randomized Study of BMS-986489 (Atigotatug + Nivolumab Fixed-dose Combination) vs Durvalumab as Consolidation Therapy Following Chemoradiotherapy in Limited-stage Small-cell Lung Cancer (TIGOS-LS)
Brief Title: BMS-986489 (Atigotatug + Nivolumab) vs Durvalumab in Limited-stage Small-cell Lung Cancer (TIGOS-LS)
Acronym: TIGOS-LS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUN 567
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Limited Stage Small Cell Lung Cancer
Keywords: limited stage small cell lung cancer; limited stage small cell lung carcinoma; LS-SCLC; Limited-stage SCLC; Nivolumab; Opdivo; fucosyl-monosialoganglioside-1; fuc-GM1; programmed cell death protein 1; PD-1 inhibitor; anti-PD-1 antibody; Durvalumab; Imfinzi; PD-L1 inhibitor; Anti-PD-L1 antibody; Limited-stage (LS)-small-cell lung cancer (SCLC); BMS-986489
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986489 (atigotatug + nivolumab) (Experimental): Participants will receive a fixed dose of BMS-986489 (atigotatug + nivolumab) intravenously each cycle. Cycles will be 28 days. Up to 125 participants will be enrolled into this arm.
  Interventions: Drug: BMS-986489
- Durvalumab (Active Comparator): Participants will receive standard of care Durvalumab intravenously each cycle. Cycles will be 28 days. Up to 125 participants will be enrolled into this arm.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: BMS-986489 — BMS-986489 (fixed dose combination of atigotatug + nivolumab) will be administered as an intravenous infusion to be given once every 4 weeks for up to 2 years.
  Arms: BMS-986489 (atigotatug + nivolumab)
Drug: Durvalumab — Durvalumab will be administered as a fixed dose intravenous infusion to be given once every 4 weeks for up to 2 years.
  Arms: Durvalumab

SUMMARY:
This is an open-label, randomized study of BMS-986489 (atigotatug + nivolumab fixed-dose combination) vs durvalumab in limited-stage (LS)-small-cell lung cancer (SCLC) participants.

The main goals of this study are to:

* Evaluate the efficacy of BMS-986489 vs durvalumab
* Evaluate the safety profile of BMS-986489

DETAILED DESCRIPTION:
This is an open-label, randomized study of BMS-986489 (atigotatug + nivolumab fixed-dose combination) vs durvalumab as consolidation therapy following chemoradiotherapy in participants with limited-stage (LS)-small-cell lung cancer (SCLC). Participants will receive concurrent chemotherapy and radiotherapy according to standard guidelines for treatment of LS-SCLC without progressive disease prior to randomization. Eligible participants will be randomly assigned to receive either BMS-986489 (atigotatug + nivolumab as a fixed-dose combination; Arm A) or durvalumab (Arm B) as consolidation therapy. Atigotatug is a first-in-class, fully human IgG1 antibody being developed for the treatment of SCLC. Atigotatug specifically binds to fuc-GM1 on the tumor cell. Nivolumab is a monoclonal anti-PD-1 antibody. Combining atigotatug with another immunotherapy may provide enhanced antitumor effects.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years-of-age at the time of signature of the Informed Consent Form (ICF)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (Appendix A)
* Histologically or cytologically confirmed pulmonary SCLC, evaluable by RECIST v1.1
* Limited-stage (LS) disease as determined by positron emission tomography (PET) scan prior to initiation of chemotherapy and radiation therapy
* Completed concurrent chemotherapy and radiotherapy for LS-SCLC without progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (computed tomography [CT] scan chest/abdomen/pelvis; Appendix B) within 42 days before date of randomization and first dose of study treatment

  * Chemotherapy should consist of a platinum and IV etoposide. Participants who received at least 3 cycles of chemotherapy will be eligible to participate.
  * Radiotherapy should be administered per institutional guidelines
* Prophylactic cranial irradiation (PCI) may be delivered at the discretion of the Investigator and institutional guidelines. PCI, if applicable, must be conducted after the end of chemoradiotherapy and completed between 14 and 42 days before date of randomization and first dose of study treatment.
* Adequate hematologic and organ function
* Willingness to abide by protocol defined contraceptive requirements for the duration of the study.

Exclusion Criteria:

* Small-cell cancer not pulmonary in origin
* Large cell neuroendocrine carcinoma
* ES-SCLC
* Mixed SCLC and NSCLC histologic features; diagnosis of NSCLC; or EGFR-activating, mutation-positive NSCLC that has transformed to SCLC
* History of severe hypersensitivity reaction to monoclonal antibodies
* Known hypersensitivity to any excipients of atigotatug, nivolumab, or durvalumab
* Grade ≥2 peripheral neuropathy by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
* Active, prior, or suspected autoimmune disease, including autoimmune neurologic disorders such as paraneoplastic syndrome involving the CNS, peripheral sensory/motor nerves, or neuromuscular junction. Exceptions to this criterion include:

  * Type 1 diabetes mellitus
  * Hypothyroidism requiring only hormone replacement
  * Skin disorders not requiring systemic treatment
  * Autoimmune conditions not expected to recur during the study
* Diseases or conditions requiring chronic systemic corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive therapy within 14 days of starting study treatment. Limited-course (<2 weeks' duration) oral steroids (10 mg prednisone or equivalent) are permitted. Bronchodilators, inhaled or topical steroids, and adrenal replacement steroid doses >10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* History of solid organ or bone marrow transplantation
* History of Grade ≥2 pneumonitis (excepting resolved infective pneumonitis)
* Any of the following cardiac criteria, currently or within the last 3 months:

  * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block, third-degree heart block, atrial fibrillation not rate controlled. Certain conditions may be considered through discussion with the Medical Monitor.
  * Congestive heart failure (New York Heart Association [NYHA] > Grade 2) or classified as Class 3 or 4 by the NYHA Functional Classification (Appendix D)
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, uncontrolled hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval (Appendix E). Certain conditions may be considered through discussion with the Medical Monitor.
  * Participants with a left ventricular ejection fraction <55% or the lower limit of normal of the institutional standard
  * Uncontrolled hypertension, defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management
  * Active coronary artery disease, including unstable or newly diagnosed angina
  * Myocardial infarction
  * History of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes)
  * History or current diagnosis of myocarditis
* As judged by the Investigator, participants with serious or uncontrolled medical disorders
* Presence of other active invasive cancers. Participants with a previously treated malignancy will be eligible to participate if treatment of that malignancy was completed at least 2 years before date of screening and the participants has no evidence of disease. Exceptions to this criterion include appropriately treated basal cell carcinoma of the skin; in situ carcinoma of uterine cervix; localized prostate cancer that has been definitively treated; or other local tumors considered cured by local treatment.
* Received sequential chemotherapy and radiotherapy as a definitive treatment for LS-SCLC
* Treatment with any of the following:

  * Any systemic anticancer chemotherapy, small molecule, biologic, or hormonal agent from a previous treatment regimen or clinical study within 21 days or 5 half-lives (whichever is longer) prior to the first dose of study treatment
  * Wide-field radiotherapy (including therapeutic radioisotopes such as strontium-89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study treatment or has not recovered from side effects of such therapy
  * Prior systemic treatment for LS-SCLC, with the exception of chemoradiotherapy and PCI
  * Prior treatment with an anti-PD-1, anti-PD-L1, anti-programmed cell death ligand 2 (anti-PD-L2), anti-CD137, anti-cytotoxic T-lymphocyte associated protein 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways
  * Prior treatment with fuc-GM-1 vaccine or targeted agent or similar vaccine targeting ganglioside antigens
  * Current treatment with immunosuppressive medications
  * Live attenuated vaccine within 100 days before first dose of study treatment
* Major surgery (excluding placement of vascular access) within 4 weeks of date of screening
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment. Note: Participants with chronic Grade 2 toxicities who are asymptomatic or adequately managed with stable medication may be eligible with approval by the Medical Monitor or Principal Investigator.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of BMS-986489 vs durvalumab by Overall Survival (OS). | From date of randomization up to 5 years. Every 8 weeks for participants who stopped treatment before disease progression and before completing 6 months of treatment and every 12 weeks for participants who stopped treatment before disease progression and
  Overall Survival (OS) is defined as the time between the date of randomization and the date of death due to any cause.

SECONDARY OUTCOMES:
Evaluate the efficacy of BMS-986489 vs durvalumab by Progression Free Survival (PFS). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Progression Free Survival (PFS) is defined as the time from start of study treatment to the date of an event, defined as the first documented radiological progression or death due to any cause.
Evaluate the efficacy of BMS-986489 vs durvalumab Objective Response Rate (ORR). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Objective Response Rate (ORR) is defined as the proportion of participants with BOR of CR or PR according to RECIST v1.1.
Evaluate the efficacy of BMS-986489 vs durvalumab by Clinical Benefit Rate (CBR). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Clinical Benefit Rate (CBR) is defined as the proportion of participants with BOR of CR or PR, or participants with SD lasting at least 180 days (i.e., ≥6 months) according to RECIST v1.1.
Evaluate the efficacy of BMS-986489 vs durvalumab by Disease Control Rate (DCR). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Disease Control Rate (DCR) is defined as the proportion of participants with BOR of CR, PR, or SD according to RECIST v1.1
Evaluate the efficacy of BMS-986489 vs durvalumab by Duration of Response (DoR). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Duration of Response (DoR) is defined as the duration from the first documented response (Complete Response (CR), Partial Response (PR), or Stable Disease (SD), according to RECIST v1.1) to the date of first documented disease progression or death.
Evaluate the efficacy of BMS-986489 vs durvalumab by Time to Progression (TtP). | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Time to Progression (TtP) is defined as the time from the date of randomization to the date of first documented disease progression, according to RECIST v1.1.
Evaluate the efficacy of BMS-986489 vs durvalumab by time to development of central nervous system (CNS) metastasis. | Every 2 cycles (8 weeks) from Cycle 1 Day 1, for the first 6 months, then every 3 cycles (12 weeks) until disease progression or death, up to 3 years. Each cycle is 28 days.
  Time to development of central nervous system (CNS) metastasis is defined as the time from the date of randomization to the date of first documented CNS metastasis.
Evaluate the number of participants with adverse events following administration of BMS-986489. | From Cycle 1 Day 1 to 100 days after the last dose of BMS-986489. Each cycle is 28 days.
  Adverse Events to be evaluated per CTCAE v5.0 criteria from first dose of BMS-986489 to 100 days after the last dose of BMS-986489.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — SCRI Development Innovations, LLC
Locations (27):
- United States (27):
  - Southern Cancer Center, Daphne, Alabama
  - Sansum Clinic, Santa Barbara, California
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Cancer Specialists - North, Orange City, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Minnesota Oncology Hematology, Maple Grove, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - White Plains Hospital Physician Associates, White Plains, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Mid Ohio Hem/ Onc dba The Mark H Zangmeister Center, Columbus, Ohio
  - Oncology Associates of Oregon (Willamette Valley Cancer Institute and Research Center), Eugene, Oregon
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology- Austin, Austin, Texas
  - Texas Oncology - Gulf Coast, Beaumont, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology - Northeast Texas, Denison, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Blue Ridge Cancer Center (Oncology & Hematology Associates of Southwest VA), Salem, Virginia

IPD SHARING:
Plan to Share IPD: No